CLINICAL TRIAL: NCT01540240
Title: Safety of Reduced Dose Zidovudine (AZT) Compared With Standard Dose AZT in Antiretroviral-naïve HIV-infected Patients: A Randomized Controlled Trial
Brief Title: Safety of Reduced Dose Zidovudine (AZT) Compared With Standard Dose AZT in Antiretroviral-naïve HIV-infected Patients
Acronym: AZTlowdose
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Rougemont Mathieu, Medical Doctor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-005
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: HIV; Zidovudine Adverse Reaction
Keywords: HIV treatment; zidovudine; dose reduction; anaemia; safety and efficacy comparison
MeSH Terms: conditions — Anemia | interventions — Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard dosage zidovudine (Active Comparator): Standard AZT arm: AZT 300 mg/3TC 150 mg(Combivir 1 cap) twice a day. Nevirapine 200 mg 1 cap twice a day.
  Interventions: Drug: Zidovudine
- low dosage zidovudine (Active Comparator)
  Interventions: Drug: Zidovudine

INTERVENTIONS:
Drug: Zidovudine — Low dosage AZT arm: AZT 200 mg/3TC 150 mg(zidovudine 100 mg 2 caps/lamivudine 150 mg 1 cap) twice a day. Nevirapine 200 mg 1 cap twice a day.
  Arms: low dosage zidovudine
Drug: Zidovudine — Standard AZT arm: AZT 300 mg/3TC 150 mg(Combivir 1 cap) twice a day. Nevirapine 200 mg 1 cap twice a day.
  Arms: standard dosage zidovudine

SUMMARY:
The primary objective of the study is to compare the tolerance and safety between a low-dose Zidovudine (AZT) containing regimen (200 mg BID) and a standard dosage (300 mg BID) in HIV patients initiating a first line antiretroviral therapy. The investigators expect that the low-dose regimen will show improved tolerability and safety compared to the standard dosage, with significant reduction in number of patients experiencing a new grade 1 to 4 anaemia or increasing their anaemia grade during the first 6 months of treatment.

The secondary objectives of the study is to compare the efficacy of the two dosing regimen, as measured by classical clinical and biological markers: the number of new AIDS defining illness, the mortality rate, the proportion of patients achieving virological success and the mean CD4 cell count increase from baseline.

DETAILED DESCRIPTION:
Existing formulations for adults include zidovudine 100mg capsule, zidovudine/3TC 300/150mg, zidovudine/3TC/NVP 300/150/200mg, zidovudine/3TC/ABC 300/150/300. Currently, international guidelines recommend a daily dose of 600 mg in 2 divided doses. Pharmacokinetic studies on zidovudine showed a twice daily regimen resulted in higher predose zidovudine-triphosphates (TP) concentrations, the active intracellular metabolite, when compared to the same daily dose given once daily. Further, a small study in Thailand study found doses of zidovudine 200 mg twice daily achieved plasma levels equivalent to the standard international 300 mg twice daily dose in individuals weighing less than 60 kg.

The clinical efficacy of zidovudine has been evaluated in randomized clinical trials using a range of doses from 300 to 1500 mg/day. In an early trial (Nordic Medical Research Councils' HIV Therapy Group 1992) comparing different dosing of zidovudine monotherapy in advanced HIV infection found no differences in death rate, or new AIDS defining events. The incidence of anaemia and leucopenia comparing 400 mg and 1200 mg daily showed a direct dose relationship: 4% to 24% (anaemia) and 3% to 22% (leucopenia) respectively. Another early trial (Fischl 1990) demonstrated an improved survival with the lower dose of zidovudine (63%) versus the high dose (52%), again with significantly more anaemia and neutropenia in the high dose zidovudine arm (p < 0.001).

High doses of zidovudine have led to increased incidence of anaemia and neutropenia, with no impairment in treatment efficacy as measured by CD4 cell count, HIV RNA level or clinical progression. In the context of new recommendations favouring the use of zidovudine over stavudine as first line treatment in resource limited settings, the investigators aim at evaluating the impact of reduced zidovudine (200 mg BID) treatment.

API (active product ingredient) production costs are the most important determinant of antiretroviral drug prices among generic manufacturers. A given percentage reduction in dosage will thus translate into a virtually equivalent percentage in drug pricing. As cART will continue to expand in Least Developed Countries, it is predicted that around 1.5 million people will take zidovudine-based regimen by 2010. Small reductions in the annual per-patient cost of AZT-based regimen could lead to significant reductions in the global cost of HIV treatment: it is estimated a 47 million US dollars savings if 9 million patients will be treated in 2014.

The present study is a prospective, randomised, 48 weeks, phase II trial. Subjects will be recruited through one site: the HIV outpatient clinic of Internal Medicine Department, CNPS Hospital, Yaoundé, Cameroun. Randomisation will be performed at initiation of ART. Patients will be randomised in one of the following treatments arms, in combination with lamivudine and an NNRTI regimen: a low-dose AZT arm (200 mg twice daily)or a standard-dose AZT arm (300 mg twice daily).

The primary endpoint is the comparison of proportions of patients experiencing a new grade 1 to 4 anaemia or increasing their anaemia grade between the two dosing AZT regimen during the first six months of treatment.

The secondary endpoints are:

* Mean haemoglobin concentration and leukocyte count changes, laboratory grade 3 and 4 adverse events rate leading or not to switch for another cART regimen.
* Differences in proportion of patients achieving virological success (VL <50 cop/ml) between the two dosing zidovudine regimen at week 24.
* Difference in proportion of patients achieving virological success ( VL <400 cop/ml) between the two dosing zidovudine regimen at week 24.
* Difference in mean viral load decline between the two groups at week 4 and 8
* Difference in mean CD4 cell count increase from baseline between the two dosing zidovudine regimen at week 8, 24.
* Difference in proportion of patients with genotype mutations in patient with detectable viral load at week 24.
* Number of new AIDS defining illness, mortality rate, drop-out rate will be compared between the two groups.

Patients will be followed individually 24 weeks for the entire period of experimental treatment. After the follow-up period, all patients included in the low dose AZT arm will be treated with standard AZT dose. They will keep their routine follow-up at the CNPS hospital.

For the first 68 patients included (half of the total cohort) in the study, the Data Safety Monitoring Board (DSMB, independently of the clinical investigators) will undergo an interim analysis at week 8 of follow-up before continuing enrollment. In this sample of patients, the efficacy of two treatment groups will be compared: an excess of 15% virological treatment failure in the low-dose AZT arm will be considered as significant. Virological treatment failure at this point is defined as a decline in viral load from baseline to the 8th week of less than 2log.

An incidence of 30% of patients experiencing new grade 1 to 4 anaemia or increasing their anaemia grade during the first 6 months of treatment is expected with the standard AZT dose regimen. A reduction of this adverse event to 10% of the patients treated by the low dose regimen would be considered as clinically significant. Thus, with a 10% of LFU expected during the follow-up period, the investigators calculate a sample size of 68 patients in each arm to detect a clinically significant difference between the two arms.

The percentage of patients experiencing a new grade 1 to 4 anaemia or increasing their anaemia grade will be compared between both treatment arms using the difference of proportion observed (Chi2 test or Fisher exact test).

The same method will be used to compare all the efficacy and safety indicators. Multivariate analysis will be used to obtain adjusted estimates of risk factors for treatment failure and for clinically significant adverse events.

Analysis on treatment safety and efficacy will be performed both in 'intention to treat" and in "per protocol".

An "intention to treat" analysis will include patients enrolled in the study who received at least one dose of study medication to which they were randomly allocated.

A "per protocol" analysis will include patients enrolled in the study who received at least one dose of study medication to which they were randomly allocated AND have reached one of the protocol defined treatment failure endpoints (death, lost to follow-up, virological failure) on the treatment they were randomly allocated or have completed the trial follow-up on the treatment they were randomly allocated.

Criteria for the termination of the trial are:

* Too low enrollment rate.
* Unsafe or unethical practices.
* Following the recommendation of the DSMB. The sponsor and investigators will ensure that this study is conducted in full compliance with the principles of the "Declaration of Helsinki" or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual. The study must fully adhere to the principles outlined in "Guideline for Good Clinical Practice" ICH Tripartite Guideline (E6, June 1996) or with local law if it affords greater protection to the subject.

This study will be conducted in accordance with the ethical principles laid out in the Declaration of Helsinki and the National Statement on Ethical Conduct in Research Involving Humans.

Investigators will obtain written informed consent from each subject participating in this study, after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study.

ELIGIBILITY:
Inclusion Criteria:

* Medical indication to initiate cART based on local guidelines
* Provision of written, informed consent
* Adults aged more than 18 years

Exclusion Criteria:

* Prior cART.
* Grade 2 to 4 baseline anaemia or leucopenia/neutropenia (WHO).
* Patients unable or unwilling to provide informed consent.
* Pregnant women
* AgHBs positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
New grade 1 to 4 anaemia or increasing anaemia grade in the two AZT dosing arms | full blood count will be assessed at week 2, week 8 and week 24 of starting antiretroviral treatment
  Differences in proportion of patients experiencing a new grade 1 to 4 anaemia or increasing their anaemia grade between the two dosing AZT regimen during the first six months of treatment. Anaemia grade will be defined by the WHO^grading of adverse events.

SECONDARY OUTCOMES:
Comparison of the immunological and virological efficacy between the two AZT dosing regimen | HIV viral load and CD4 cell count will be assessed at week 4, week 8 and week 24 of starting antiretroviral treatment
  The efficacy of the two dosing regimen will be measured by: the number of new AIDS defining illness, the mortality rate, the proportion of patients achieving virological success and the mean CD4 cell count increase from baseline. Secondary variables that will compare the efficacy and safety of the two AZT dosing regimen are: the viral load decrease in log after at week 4 and 8, the proportion of patients below 50 copies/ml at week 24, the proportion of patients below 400 cop/ml at week 24, the proportion of patients experiencing anaemia and neutropenia grade 3 and 4 at week 4, 8 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Peter N Ngang, MD, Principal Investigator — CNPS hospital, Yaoundé, Cameroun
Locations (1):
- CNPS Hospital, Yaoundé, Cameroon